CLINICAL TRIAL: NCT05158023
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Dose-Ranging Trial to Evaluate the Efficacy and Safety of ASLAN004 in Adult Patients With Moderate-to-Severe Atopic Dermatitis
Brief Title: Phase 2b Study of ASLAN004 in Adults With Moderate-to-Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ASLAN Pharmaceuticals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASLAN004-003
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; IL-13; ASLAN004; IL-13Rα1; Eczema; Anti-IL-13Rα1; atopic eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo every two weeks q2w (Placebo Comparator): Placebo q2w - placebo loading dose equivalents at Baseline and Week 1, then placebo dose equivalents every 2 weeks (q2w) from Week 2 to Week 14.
  Interventions: Drug: Placebo Comparator
- ASLAN004 300 mg q2w (Experimental): ASLAN004 300 mg q2w - loading doses at Baseline and Week 1, followed by regular doses of 300mg q2w from Week 2 to Week 14.
  Interventions: Biological: ASLAN004
- ASLAN004 400 mg q2w (Experimental): ASLAN004 400 mg q2w - loading doses at Baseline, Week 1 and Week 2, followed by regular doses of 400 mg ASLAN004, alternating with placebo dose equivalents, q2W from Week 4 to Week 14.
  Interventions: Biological: ASLAN004
- ASLAN004 400 mg every four weeks q4w (Experimental): ASLAN004 400 mg q4w - loading doses at Baseline, Week 1 and Week 2, followed by regular doses of 400 mg or alternating placebo (q2W) to Week 14.
  Interventions: Biological: ASLAN004
- ASLAN004 600 mg q4w (Experimental): ASLAN004 600 mg q4w - loading doses at Baseline, Week 1 and Week 2, followed by regular doses of 600 mg ASLAN004, alternating with placebo dose equivalents, q2W from Week 4 to Week 14.
  Interventions: Biological: ASLAN004

INTERVENTIONS:
Drug: Placebo Comparator — Sterile solution for subcutaneous injection
  Arms: Placebo every two weeks q2w
Biological: ASLAN004 — Sterile solution for subcutaneous injection
  Arms: ASLAN004 300 mg q2w
Biological: ASLAN004 — Sterile solution for subcutaneous injection
  Arms: ASLAN004 400 mg q2w
Biological: ASLAN004 — Sterile solution for subcutaneous injection
  Arms: ASLAN004 400 mg every four weeks q4w
Biological: ASLAN004 — Sterile solution for subcutaneous injection
  Arms: ASLAN004 600 mg q4w

SUMMARY:
Phase 2b study designed to evaluate the efficacy and safety of ASLAN004 in adult patients with moderate-to-severe Atopic Dermatitis (AD) who are candidates for systemic therapy. This study will have 5 treatment arms (4 active and 1 placebo).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients with a clinical diagnosis of AD for at least 1 year;
2. vIGA score of ≥3 at Screening and Baseline;
3. ≥10% BSA of AD involvement at Screening and Baseline;
4. EASI score ≥16 at Screening and Baseline;
5. History of inadequate response to treatment with topical corticosteroids (TCS) or topical calcineurin inhibitors (TCI);
6. Twice daily application of a consistent amount of topical emollient for at least 7 days prior to randomization.

Exclusion Criteria:

1. Immunosuppressive/immunomodulating drugs, systemic therapies or phototherapy within 4 weeks prior to randomization;
2. Treatment with leukotriene inhibitors within 4 weeks prior to randomization;
3. Treatment with topical therapies (including TCS, TCI, topical phosphodiesterase inhibitors, topical JAK inhibitors) or prescription moisturizers, within 1 week prior to randomization;
4. Previous treatment at any time prior to randomization with monoclonal antibody / biologic therapeutic agents as follows;

   1. Prior exposure to dupilumab (Dupixent®) which was discontinued due to lack of efficacy, loss of response, or adverse event;
   2. Investigational or approved agents targeting interleukins IL-4 or IL-13 ligands or receptors of IL-4 or IL-13, including but not limited to lebrikizumab, tralokinumab or ASLAN004;
   3. Other investigational or approved biologic drug within 16 weeks or within 5 half-lives (if known), whichever is longer, prior to the Baseline visit;
   4. Cell-depleting biologics, including, but not limited to, rituximab within 6 months prior to the Baseline visit;
5. Inadequate organ function, abnormal lab result, uncontrolled blood pressure or other health condition considered clinically significant by the investigator at the Screening visit;
6. History of HIV, Hepatitis B, Hepatitis C or active/latent Tuberculosis infection;
7. History of immunosuppression including history of invasive opportunistic infections;
8. Treatment with live attenuated vaccine within 8 weeks prior to randomization;
9. Parasitic infection within 4 weeks prior to baseline travel within 3 months prior to randomization to areas of high parasitic exposure;
10. Have skin comorbidities that in the opinion of the Investigator may interfere with study assessments;
11. Pregnant or breastfeeding women;
12. Patients unwilling to use adequate birth control.
13. Active COVID infection at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
Percent change from Baseline in Eczema Area and Severity Index (EASI) at Week 16 | Baseline, Week 16
  The EASI score is used to measure the severity and extent of AD and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD

SECONDARY OUTCOMES:
Proportion of patients achieving validated Investigator's Global Assessment (vIGA) response of 0 (clear) or 1 (almost clear) at Week 16 | Week 16
  IGA is an assessment scale used to determine severity of AD and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response is an IGA score of 0 (clear) or 1 (almost clear).
Proportion of patients with EASI 50, 75 and 90 at Week 16 | Week 16
  EASI scores range from 0 to 72 (severe)The EASI responder is defined as a participant who achieves a ≥50% improvement (EASI 50), ≥75% improvement (EASI 75), or ≥90% improvement (EASI 90) from baseline in the EASI score.
Proportion of patients with EASI <7 at Week 16 | Week 16
  EASI scores range from 0 to 72 (severe)
Percent Change in EASI score from Baseline over time | Baseline, Week 16
  EASI scores range from 0 to 72 (severe)
Absolute and percent change in Pruritus Numerical Rating Scale (P-NRS) over time | Baseline, Week 16
  The P-NRS is an 11-point scale used by patients to assess their worst itch severity over the past 24 hours, with 0 indicating no itch and 10 indicating the worst itch imaginable. Pruritus assessments will be recorded daily by the patient using an electronic diary
Proportion of patients achieving a 4-point reduction in P-NRS | Baseline, Week 16
  The P-NRS is an 11-point scale used by patients to assess their worst itch severity over the past 24 hours, with 0 indicating no itch and 10 indicating the worst itch imaginable. Pruritus assessments will be recorded daily by the patient using an electronic diary.
Change in Body Surface Area (BSA) affected with AD | Baseline, Week 16
  BSA ranges from 0% to 100 % with higher values representing greater extent of AD.
Change in SCORing Atopic Dermatitis (SCORAD) from Baseline to Week 16 | Baseline, Week 16
  The SCORAD is a validated measure of the extent and severity of atopic dermatitis lesions, along with subjective symptoms. The score ranges from 0 to 103, with higher values indicating a more extensive and/or severe condition.
Change in Dermatology Life Quality Index (DLQI) from Baseline to Week 16 | Baseline, Week 16
  The DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the patient's perception of the impact of AD disease symptoms and treatment on their quality of life (QoL). The 10 questions assess QoL over the past week, with an overall scoring of 0 (absent disease) to 30 (severe disease). A high score is indicative of a poor QoL.
Change in Patient-Oriented Eczema Measure (POEM) from Baseline to Week 16 | Baseline to Week 16
  The POEM is a 7-item questionnaire that assesses disease symptoms (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) with a scoring system of 0 (absent disease) to 28 (severe disease) (high score indicative of poor quality of life [QOL])
Change in the European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) Index Score United States and United Kingdom Algorithm from Baseline to Week 16 | Baseline, Week 16
  The EQ-5D-5L is a 2-part measurement. The second part is assessed using a VAS that ranges from 0 to 100 millimeter (mm), where 0 is the worst health you can imagine and 100 is the best health you can imagine
Change in Hospital Anxiety Depression Scale (HADS) from Baseline to Week 16 | Baseline to Week 16
  HADS is a 14-item scale. Seven of the items relate to anxiety and seven items relate to depression. Each item on the questionnaire is scored from 0 (minimum score) - 3 (maximum score) and this means that a person can score between 0 (no symptoms) and 21 (severe symptoms) for either anxiety or depression. The total HADS score or subscores may be regarded as a global measure of psychological distress; higher scores indicate greater levels of anxiety or depression.
Absolute and percent change in sleep disturbance SD-NRS over time | Baseline to Week 16
  The SD-NRS is an 11-point scale used by patients to assess their sleep disturbance severity over the past 24 hours, with 0 indicating no or minimal sleep disturbance and 10 indicating the worst imaginable sleep disturbance. SD-NRS assessments will be recorded daily by the patient using an electronic diary.
Proportion of patients achieving a 4-point reduction in SD-NRS from Baseline to at Week 16 | Baseline to Week 16
Number of Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs) from study drug administration (Day 1) to Week 28 | : Baseline to Week 28
  TEAEs are defined as AEs that develop or worsen or become serious during on-treatment period (time from the first dose of study drug until Week 28. A TESAE is defined as any untoward medical occurrence that results in any of the following outcomes: death, life-threatening, requires initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or is considered as medically important event. Any TEAE includes participants with both serious and non-serious AEs.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — ASLAN Pharmaceuticals
Locations (78):
- United States (45):
  - ASLAN Investigative Site, Birmingham, Alabama
  - ASLAN Investigative Site, Little Rock, Arkansas
  - Tooraj Raoof, MD, Encino, California
  - ASLAN Investigative Site, Fountain Valley, California
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - ASLAN Investigative Site, Los Angeles, California
  - MedDerm Associates, San Diego, California
  - Clinical Science Institute, Santa Monica, California
  - Skin Care Research, LLC, Boca Raton, Florida
  - Encore Medical Research of Boynton Beach, Boynton Beach, Florida
  - Driven Research, LLC, Coral Gables, Florida
  - Aby's New Generation Research, Inc., Hialeah, Florida
  - ASLAN Investigative Site, Hollywood, Florida
  - Skin Research of South Florida, Miami, Florida
  - ASLAN Investigative Site, Miami, Florida
  - ASLAN Investigative Site, North Miami Beach, Florida
  - ASLAN Investigative Site, Saint Augustine, Florida
  - ASLAN Investigative Site, Tampa, Florida
  - ForCare Clinical Research, Tampa, Florida
  - ASLAN Investigative Site, Columbus, Georgia
  - Skin Care Physicians of Georgia, Macon, Georgia
  - ASLAN Investigative Site, Meridian, Idaho
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - ASLAN Investigative Site, Louisville, Kentucky
  - ASLAN Investigative Site, Baton Rouge, Louisiana
  - Allcutis Research LLC, Beverly, Massachusetts
  - ASLAN Investigative Site, Quincy, Massachusetts
  - ASLAN Investigative Site, Ann Arbor, Michigan
  - ASLAN Investigative Site, Las Vegas, Nevada
  - Forest Hills Dermatology Group, Kew Gardens, New York
  - Bobby Buka MD, PC, New York, New York
  - ASLAN Investigative Site, New York, New York
  - ASLAN Investigative Site, Medford, Oregon
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Clinical Research Center of the Carolinas, Charleston, South Carolina
  - ASLAN Investigative Sites, Rapid City, South Dakota
  - ASLAN Investigative Site, Nashville, Tennessee
  - Dermatology Treatment and Research Center, Dallas, Texas
  - Modern Research Associates, Dallas, Texas
  - Menter Dermatology Research Institute, Dallas, Texas
  - Center for Clinical Studies LTD, LLP, Houston, Texas
  - ASLAN Investigative Site, San Antonio, Texas
  - ASLAN Investigative Site, South Jordan, Utah
- Australia (6):
  - Premier Specialist, Kogarah, New South Wales
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - Veracity Clinical Research, Woolloongabba, Queensland
  - Eastern Clinical Research, Box Hill, Victoria
  - Skin Health Institute, Carlton, Victoria
  - Fremantle Dermatology, Fremantle, Western Australia
- Canada (7):
  - Wiseman Dermatology Research, Inc., Winnipeg, Manitoba
  - DermEffects, London, Ontario
  - ASLAN Investigative Site, Markham, Ontario
  - Gordon Sussman Clinical Research Inc., North York, Ontario
  - Skin Centre for Dermatology, Peterborough, Ontario
  - Centre de Recherche Saint-Louis (Quebec), Québec, Quebec
  - Centre de Recherche dermatologique du Quebec Metropolitain, Québec, Quebec
- ASLAN Investigative Site, Santo Domingo, Dominican Republic
- India (8):
  - B. J. Medical College and Civic Hospital, Asarwa, Ahmedabad
  - Nirmal Hospital Pvt Ltd., Surat, Gujarat
  - NKP Salve Institute of Medical Sciences & Research Centre and Lata Mangeshkar Hospital, Nagpur, Maharashtra
  - D Y Patil Hospital, Navi Mumbai, Maharashtra
  - Calcutta School of Tropical Medicine, Kolkata, West Bengal
  - Sir Ganga Ram Hospital, New Delhi
  - Lifepoint Multispeciality Hospital, Pune
  - King George Hospital, Visakhapatnam
- Clinical Trials NZ, Hamilton, New Zealand
- Poland (7):
  - ASLAN Investigative Site, Bydgoszcz
  - ASLAN Investigative Site, Katowice
  - ASLAN Investigative Site, Krakow
  - ASLAN Investigative Site, Lodz
  - ASLAN Investigative Site, Tarnów
  - ASLAN Investigative Site, Warsaw
  - ASLAN Investigative Site, Wroclaw
- Singapore (3):
  - ASLAN Investigative Site, Singapore
  - KK Women's and Children's Hospital, Singapore
  - National Skin Centre, Singapore

IPD SHARING:
Plan to Share IPD: No